CLINICAL TRIAL: NCT03722966
Title: A Comparison of the Effectiveness of Combination Varenicline and Oral Nicotine Replacement Therapy Versus Varenicline Alone for Smoking Cessation: a Pilot Study
Brief Title: Effectiveness of Combination Varenicline and Oral Nicotine Replacement Therapy (COMBO)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following the Chantix recall, Pfizer stopped providing medication for the study and and new study enrollments were discontinued.
Sponsor: University of Oklahoma (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10184
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; varenicline; nicotine gum; nicotine lozenges; nicotine replacement therapy; adherence; mHealth
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Nicotine Replacement Therapy; Nicotine Chewing Gum; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Varenicline/Counseling + Med Reminders (VAR+REM) (Experimental): Participants will receive behavioral tobacco cessation counseling, a 13-week course of varenicline, and automated medication reminders via their smartphones.
  Interventions: Drug: Varenicline; Behavioral: Medication Reminders; Behavioral: Tobacco Cessation Counseling
- Varenicline/Counseling (VAR+NREM) (Experimental): Participants will receive behavioral tobacco cessation counseling, a 13-week course of varenicline, and no automated medication reminders.
  Interventions: Drug: Varenicline; Behavioral: Tobacco Cessation Counseling
- Varenicline/Counseling + Oral NRT (VAR+NRT+NREM) (Experimental): Participants will receive behavioral tobacco cessation counseling, a 13-week course of varenicline, 12 weeks of oral nicotine replacement therapy (NRT; gum or lozenge), and no automated medication reminders.
  Interventions: Drug: Varenicline; Drug: Oral Nicotine Replacement Therapy (NRT); Behavioral: Tobacco Cessation Counseling
- Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM) (Experimental): Participants will receive behavioral tobacco cessation counseling, a 13-week course of varenicline, 12 weeks of oral nicotine replacement therapy (NRT; gum or lozenge), and automated medication reminders via their smartphones.
  Interventions: Drug: Varenicline; Drug: Oral Nicotine Replacement Therapy (NRT); Behavioral: Medication Reminders; Behavioral: Tobacco Cessation Counseling

INTERVENTIONS:
Drug: Varenicline — All participants will be offered a 13-week course of varenicline (including a 1 week titration period). Dosage and administration per manufacturer: 0.5mg once daily for days 1-3 and 0.5mg twice daily for days 4-7 encompass the titration period, then 1mg twice daily for 12 weeks. An additional 12 weeks of treatment is recommended for long-term abstinence.
  Other Names: Chantix
Drug: Oral Nicotine Replacement Therapy (NRT) — Half of study participants will be randomly assigned to receive oral nicotine replacement therapy (4mg gum or 4mg lozenge, depending on preference; to be used every 1-2 hours as urges occur) in addition to varenicline.
  Other Names: Nicotine Gum (4mg); Nicotine Lozenge (4mg)
  Arms: Varenicline/Counseling + Oral NRT (VAR+NRT+NREM); Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Behavioral: Medication Reminders — Half of study participants will be randomly assigned to receive automated medication reminders via their smartphones.
  Arms: Varenicline/Counseling + Med Reminders (VAR+REM); Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Behavioral: Tobacco Cessation Counseling — All participants will be offered 6 weekly tobacco cessation counseling sessions with a Tobacco Treatment Specialist.

SUMMARY:
Varenicline is considered to be a first-line tobacco cessation treatment. Previous studies have evaluated the impact of the combination of varenicline and nicotine patches (versus varenicline alone) on smoking cessation, though findings have been equivocal. No studies to date have evaluated the combination of varenicline and oral nicotine replacement therapy (NRT; i.e., nicotine lozenges or gum). Nicotine lozenges and gum can provide acute relief during cravings and high risk situations, which offers individuals the flexibility to deliver nicotine when they need it most (in contrast with the continuous and passive delivery of nicotine offered via the patch). Prospective clinical trials are needed in real-world settings to determine whether the combination of varenicline and oral nicotine replacement therapy (i.e., lozenges, gum) is superior to varenicline alone for smoking cessation. The proposed pilot randomized trial would enroll 100 participants over 1 year (≈8 participants per month) utilizing a 2x2 factorial design. Twelve weeks of a pharmacological intervention [varenicline + oral NRT (VAR+N) vs. varenicline alone (VAR)] will be crossed with automated medication reminders (reminder messages vs. no reminder messages). All participants will receive an adapted version of the standard counseling offered through the Tobacco Treatment Research Program (TTRP).

The primary outcomes will be biochemically-verified smoking cessation at 12 and 26 weeks following a scheduled quit attempt (1 week after enrollment). Smartphone-based ecological momentary assessment (EMA) will be employed to measure withdrawal symptoms, medication adherence, side effects, and adverse events using the Insight™ platform developed by the Stephenson Cancer Center (SCC) mHealth Shared Resource. This pilot study will provide information regarding the feasibility, acceptability, and preliminary efficacy of combination varenicline and oral NRT for smoking cessation, which will support an NIH funding application for a larger, adequately powered study.

DETAILED DESCRIPTION:
Tobacco Treatment Research Program (TTRP).The TTRP led by Dr. Darla Kendzor and located at the University of Oklahoma Health Science Center (OUHSC), offers free tobacco cessation treatment to adults from campus or the community who would like to quit using tobacco. The proposed study would take place within the context of the TTRP. Individuals are linked with the TTRP via the electronic medical record and 1-click referrals from clinical departments at the OUHSC or SCC; or from the community by phone [(405) 271-QUIT (7848)], email (ttrp@ouhsc.edu), or fax referrals. Treatment includes counseling with a Tobacco Treatment Specialist either in-person or over the telephone and pharmacological treatment.

Baseline (1-Week Pre-quit; Visit 1):

Informed Consent/Screening. Informed consent will be obtained from all participants in a private room in the TTRP. Individuals will be included in the study if they: 1) are ≥ 18 years of age, 2) demonstrate > 6th grade English literacy level, 3) agree to install the study smartphone application onto their personal phone (or agree to carry a study-provided phone with the app), 4) agree to complete phone-based or in-person surveys through 26 weeks post-quit date, 5) have an expired CO level > 7 ppm at the baseline screening visit suggestive of current smoking, 6) currently smoke ≥ 5 cigarettes per day, 7) are willing to initiate a quit attempt 7 days after the baseline visit (enrollment). Individuals will be excluded from the study if they 1) have a history of seizures or allergic reaction to varenicline, 2) report current suicidality, 3) are taking anti-depressant or anti-psychotic medications, or 4) are pregnant, planning to become pregnant, or currently breastfeeding. Please note that the smartphone application used in this pilot study is only available in English.

Smartphones. Participants will be guided through the process of downloading the InsightTM smartphone application onto their personal smartphone and they will be asked to complete daily EMAs during the 12 week period when they are taking their study medication(s). Those who do not possess a phone that meets the minimum requirements to download the Insight™ app, will be provided with a study phone. The smartphone app home screen will include: 1) a "Call Staff" function/button that automatically calls study staff when participants have problems with the app, and 2) a "Payment" function/button that enables participants to track their current level of compliance with phone-based surveys and level of compensation. At the baseline visit, all participants will receive training about how to use the smartphone app to complete EMA and how to use the "Call Staff" and "Payment" button/options. Participants will be instructed to quit smoking at bedtime or 10:00 pm (whichever occurs first), 6 days following their Baseline session. The app will remind participants about their approaching quit date during each day of the pre-cessation period.

Questionnaires and Other Measures. Participants will complete self-report questionnaires on a tablet computer; and expired CO, weight, and height will be measured in a private room to ensure confidentiality.

Varenicline. All participants will be evaluated by the study physician, and prescribed varenicline (if eligible). Individuals with a history of seizures, allergic reaction to varenicline, and/or those who are pregnant, planning to become pregnant, or breastfeeding will be excluded from the proposed study. As a precaution, individuals who report current cardiovascular disease will require clearance from the study physician or their personal physician to use varenicline. Notably, recent research has indicated that neither varenicline nor NRT increases the risk of serious cardiovascular events. In December 2016, the FDA lifted the boxed warning for varenicline after findings were published from a large clinical trial showing that the risk of neuropsychiatric adverse events associated with varenicline did not differ from the nicotine patch or placebo, and that varenicline was more effective for smoking cessation than the nicotine patch, bupropion, and placebo (the nicotine patch and bupropion were more effective than placebo). Participants will be excluded for current suicidality and current use of anti-depressant and anti-psychotic medications, which are suggestive of severe and/or unstable mental illness. As a precaution, female participants will be advised to avoid pregnancy while taking varenicline and to discontinue the medication should they become pregnant. However, the findings of observational research suggests that taking varenicline does not appear to be harmful during pregnancy. During the first (pre-quit) week of the study, participants will continue smoking and begin taking varenicline. Doses are titrated during the first week of medication (days 1-3: 0.5 mg once daily; days 4-7: 0.5 mg twice daily).

Oral NRT. Participants randomized to VAR+N will be provided with a supply of 4 mg nicotine lozenges or 4 mg gum (depending on participant preference) and instructed to use a piece every 1-2 hours (12-24 per day) after they quit smoking, and especially when they have the urge to smoke.

Developing a Quit Plan. Eligible participants will meet with a tobacco cessation counselor who will provide an overview of the tobacco cessation program, and help participants to set and prepare for their quit date. Participants will be asked to quit smoking the evening prior to their next weekly appointment.

Randomization. At the conclusion of the first visit, participants will be randomized to one of the four cells within the 2x2 factorial design: pharmacological treatment (VAR+N vs. VAR) and medication reminders (reminders vs. no reminders) at the baseline visit. Adaptive randomization will be used to assign participants to groups based upon race, sex, cigarettes smoked per day, and education.

Quit Day (Visit 2; 1-Week Post-Enrollment):

Questionnaires and Other Measures. Participants will complete self-report questionnaires on a tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality.

Oral NRT. Participants randomized to VAR+N will be instructed to use a piece of gum or lozenge at least every 1-2 hours (12-24 per day), and especially when they have the urge to smoke. Participants assigned to VAR+N with medication reminders will receive smartphone prompts (through the Insight™ app) every 2 hours (during waking hours) reminding them to use a piece of gum or a lozenge when they have cravings and at least every 1-2 hours.

Counseling. Participants will complete an in-person counseling session with a Tobacco Treatment Specialist. Since participants were scheduled to quit smoking the evening prior, the counselor will check in with participants about the difficulties and successes they have experienced, and plan for any challenging situations that are anticipated. Advice and support will be provided as needed.

Weekly Telephone Counseling Sessions (1, 2, and, 3 weeks post-quit) Following the quit day, 3 additional weekly telephone counseling sessions will be scheduled. Topics will include 1) the impact of tobacco on health/benefits of quitting, 2) stress management strategies, 3) making positive lifestyle changes, 4) developing coping skills, and 5) relapse prevention. The counselor will check in with participants each week about the difficulties and successes they have experienced, and plan for any challenging situations that are anticipated. Advice and support will be provided as needed. Participants will be reminded to take their varenicline dose twice daily (VAR+N and VAR), and to use a piece of gum or a lozenge at least every 1-2 hours (VAR+N only) and especially when they have the urge to smoke.

4-Weeks Post-Quit Day (Visit 3):

Questionnaires and Other Measures. Participants will complete self-report questionnaires on a tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality.

Oral NRT. Participants randomized to VAR+N will be instructed to continue using a piece of gum or lozenge every 1-2 hours (12-24 per day), and to begin reducing to at least every 2-4 hours (6-12 per day). Additional supply of gum or lozenges will be provided at this visit. VAR+N participants will receive a smartphone reminder prompt to use a piece of gum or lozenge every 2 hours during waking hours through 6 weeks post-quit, and every 4 hours during post-quit weeks 7-12.

Counseling. Participants will complete an in-person counseling session with a Tobacco Treatment Specialist. The counselor will check in with participants each week about the difficulties and successes they have experienced, and plan for any challenging situations that are anticipated. Advice and support will be provided as needed.

8-Weeks Post-Quit Day (Visit 4):

Questionnaires and Other Measures. Participants will complete self-report questionnaires on a tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality.

Oral NRT. Participants randomized to VAR+N will be instructed to continue using a piece of gum or lozenge every 2-4 hours (6-12 per day), and to begin reducing to at least every 4-8 hours (3-6 per day). Additional supply of gum or lozenges will be provided at this visit. VAR+N participants will receive a smartphone prompt every 4 hours (during waking hours) through 12 weeks post-quit reminding them to use a piece of gum or a lozenge as directed.

12-Weeks Post-Quit Day (Visit 5):

Questionnaires and Other Measures. Participants will complete self-report questionnaires on a tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will be asked to return their study-provided smartphones after they have completed their 12 week course of varenicline.

Oral NRT. Participants randomized to VAR+N will be asked to discontinue using oral NRT.

26-Weeks Post-Quit Day (Visit 6):

Questionnaires and Other Measures. Participants will complete self-report questionnaires on a tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* ≥ 6th grade English literacy
* agree to use personal or study-provided smartphone/applications
* agree to complete phone-based or in-person surveys throughout 26 week study
* expired CO > 6 ppm at baseline visit (suggesting current smoker)
* currently smoke ≥ 5 cigarettes per day
* willing to make quit attempt 7 days after baseline visit

Exclusion Criteria:

* < 18 years of age
* history of seizures or allergic reaction to varenicline
* report current suicidality
* taking anti-depressants or anti-psychotic medications
* pregnant or planning to become pregnant
* currently breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla Kendzor, PhD, Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sifat M, Hebert ET, Ahluwalia JS, Businelle MS, Waring JJC, Frank-Pearce SG, Bryer C, Benson L, Madison S, Planas LG, Baranskaya I, Kendzor DE. Varenicline Combined With Oral Nicotine Replacement Therapy and Smartphone-Based Medication Reminders for Smoking Cessation: Feasibility Randomized Controlled Trial. JMIR Form Res. 2023 Oct 27;7:e48857. doi: 10.2196/48857. PMID 37889541
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline/Counseling + No Reminders (VAR+NREM): Participants will receive behavioral tobacco cessation counseling, a 13-week course of varenicline, and no automated medication reminders.
  Varenicline: All participants will be offered a 13-week course of varenicline (including a 1 week titration period). Dosage and administration per manufacturer: 0.5mg once daily for days 1-3 and 0.5mg twice daily for days 4-7 encompass the titration period, then 1mg twice daily for 12 weeks. An additional 12 weeks of treatment is recommended for long-term abstinence.
  Tobacco Cessation Counseling: All participants will be offered 6 weekly tobacco cessation counseling sessions with a Tobacco Treatment Specialist.
- Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM): Participants will receive behavioral tobacco cessation counseling, a 13-week course of varenicline, 12 weeks of oral nicotine replacement therapy (NRT; gum or lozenge), and no automated medication reminders.
  Varenicline: All participants will be offered a 13-week course of varenicline (including a 1 week titration period). Dosage and administration per manufacturer: 0.5mg once daily for days 1-3 and 0.5mg twice daily for days 4-7 encompass the titration period, then 1mg twice daily for 12 weeks. An additional 12 weeks of treatment is recommended for long-term abstinence.
  Oral Nicotine Replacement Therapy (NRT): Half of study participants will be randomly assigned to receive oral nicotine replacement therapy (4mg gum or 4mg lozenge, depending on preference; to be used every 1-2 hours as urges occur) in addition to varenicline.
  Tobacco Cessation Counseling: All participants will be offered 6 weekly tobacco cessation counseling sessions with a Tobacco Treatment Specialist.
Period: Overall Study
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling + No Reminders (VAR+NREM) | Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Started | 2 | 12 | 11 | 9
Completed | 1 | 9 | 7 | 7
Not Completed | 1 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling + No Reminders (VAR+NREM) | Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM) | Total
Number analyzed (Participants) | 2 | 12 | 11 | 9 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (4.950) | 50.75 (9.016) | 56.36 (9.102) | 54.56 (10.608) | 54.15 (9.410)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 5 | 4 | 17
  Male | 1 | 5 | 6 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 0 | 5
  White | 2 | 6 | 8 | 8 | 24
  More than one race | 0 | 2 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 12 | 11 | 9 | 34
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: Cigarettes per day] | 17.50 (10.607) | 16.42 (5.316) | 20.27 (11.429) | 21.11 (10.105) | 18.97 (9.027)

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-Verified Smoking Cessation
Description: Self-reported abstinence over the prior 7-days with a carbon monoxide value <7 ppm (in exhaled breath) at 12 weeks post-quit date
Time Frame: 12 weeks post-quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling + No Reminders (VAR+NREM) | Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Number analyzed (Participants) | 2 | 12 | 11 | 9
Participants | 1 | 2 | 1 | 5

2. Primary Outcome: Biochemically-Verified Smoking Cessation
Description: Self-reported abstinence over the prior 7-days in conjunction with a carbon monoxide value <7 ppm (in exhaled breath) at 26 weeks post-quit date
Time Frame: 26 weeks post-quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling + No Reminders (VAR+NREM) | Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Number analyzed (Participants) | 2 | 12 | 11 | 9
Participants | 0 | 0 | 2 | 2

3. Secondary Outcome: Varenicline Adherence
Description: Total number of days of complete varenicline adherence from 1-week pre-quit through 12 weeks post-quit (91 days possible). Complete varenicline adherence was indicated when participants reported taking varenicline daily as prescribed.
Time Frame: 1 week pre-quit though 12 weeks following a scheduled quit date (13 weeks)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling + No Reminders (VAR+NREM) | Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Number analyzed (Participants) | 2 | 12 | 11 | 9
Days | 81.50 (0.71) | 45.58 (30.44) | 35.00 (34.74) | 53.44 (31.22)

4. Secondary Outcome: Oral NRT Adherence
Description: Average daily pieces of gum/lozenges used over the first 12 weeks following a scheduled quit date.
Time Frame: 12 weeks post-quit date
Population: Participants in the VAR+ REM and VAR+NREM groups did not receive oral NRT and therefore do not have values.
Measure: Mean (Standard Deviation); unit: Daily pieces of NRT used
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling + No Reminders (VAR+NREM) | Varenicline/Counseling + Oral NRT + No Reminders (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
Number analyzed (Participants) | 0 | 0 | 9 | 9
Daily pieces of NRT used |  |  | 7.44 (9.80) | 14.00 (15.57)

ADVERSE EVENTS:
Time Frame: 27 weeks (1-week pre-quit through 26 weeks post-quit)
Arm/Group | Varenicline/Counseling + Med Reminders (VAR+REM) | Varenicline/Counseling (VAR+NREM) | Varenicline/Counseling + Oral NRT (VAR+NRT+NREM) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/12 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/12 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/2 | 3/12 | 3/11 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline/Counseling + Med Reminders (VAR+REM) (N=2) | Varenicline/Counseling (VAR+NREM) (N=12) | Varenicline/Counseling + Oral NRT (VAR+NRT+NREM) (N=11) | Varenicline/Counseling + Oral NRT + Med Reminders (VAR+NRT+REM) (N=9)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (5) | 3 (8) — Score >=5 on the Patient Health Questionnaire Depression (PHQ)-9
Sleep Problems (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Nausea with or without vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was discontinued early due to the recall of varenicline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT03722966/Prot_SAP_000.pdf